CLINICAL TRIAL: NCT02689271
Title: CombIning advaNces in imagiNg With biOmarkers for improVed Diagnosis of Aggressive prosTate cancEr
Acronym: INNOVATE
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 15/0692
Record Dates: First submitted 2016-02-12; First posted 2016-02-23 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Prostate Cancer
Keywords: MRI; Magnetic resonance imaging; Biomarkers; Fluidics; Diffusion MRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MRI — VERDICT diffusion-weighted microstructure imaging sequence

SUMMARY:
To enable the paradigm of mp-MRI before biopsy in all patients with suspected prostate cancer by better selecting patients who will benefit from diagnostic MRI and by improving the performance of the mp-MRI itself

DETAILED DESCRIPTION:
Patients will undergo an advanced diffusion-weighted MRI sequence called VERDICT with the intention of better characterising prostate cancer. A panel of serum and urine biomarkers will also be analysed, which we hope will predict those patients who go on have a positive MRI.

OBJECTIVES:

* To establish a fluidic marker - prostate MRI paradigm which: (i) utilises fluidic markers to rationalise selection of patients with significant prostate cancer; and (ii) improves the diagnostic accuracy of imaging over and above standard multiparametric (mp) MRI
* Enable a pathway for rapid clinical evaluation of emerging fluidic markers and exosomes
* Assess the repeatability of VERDICT MRI
* Ascertain whether VERDICT derived quantitative parameters correlate with quantitative histological parameters
* Develop a database of fluidic marker and VERDICT characterised, mp-MRI, histologically validated patients for subsequent exploratory and longitudinal outcome analysis

ELIGIBILITY:
Inclusion Criteria:

* Men referred to University College London Hospital (UCLH) for prostate mp-MRI following biopsy elsewhere and biopsy naive men presenting to UCLH with a clinical suspicion of prostate cancer.

Exclusion Criteria:

* Men unable to have a MRI scan, or in whom artefact would reduce quality of MRI
* Men unable to given informed consent
* Previous treatment (prostatectomy, radiotherapy, brachytherapy) of prostate cancer
* On-going hormonal treatment for prostate cancer
* Previous biopsy within 6 months of scheduled mp-MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with suspected prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of VERDICT MRI | 3 - 6 months (after targeted biopsy or follow up MRI)
  Radiological assessment with added VERDICT MRI improves the specificity of mp-MRI for detection of significant prostate cancer by >10% above standard multi-parametric MRI alone.

CONTACTS AND LOCATIONS:
Locations (1):
- University College London Hospital, Camden, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Rogers H, Kanber B, Clemente J, Pye H, Johnston EW, Parry T, Grey A, Dinneen E, Shaw G, Heavey S, Stopka-Farooqui U, Haider A, Freeman A, Giganti F, Atkinson D, Moore CM, Whitaker HC, Alexander DC, Panagiotaki E, Punwani S. Avoiding Unnecessary Biopsy after Multiparametric Prostate MRI with VERDICT Analysis: The INNOVATE Study. Radiology. 2022 Dec;305(3):623-630. doi: 10.1148/radiol.212536. Epub 2022 Aug 2. PMID 35916679
- [Derived] Johnston E, Pye H, Bonet-Carne E, Panagiotaki E, Patel D, Galazi M, Heavey S, Carmona L, Freeman A, Trevisan G, Allen C, Kirkham A, Burling K, Stevens N, Hawkes D, Emberton M, Moore C, Ahmed HU, Atkinson D, Rodriguez-Justo M, Ng T, Alexander D, Whitaker H, Punwani S. INNOVATE: A prospective cohort study combining serum and urinary biomarkers with novel diffusion-weighted magnetic resonance imaging for the prediction and characterization of prostate cancer. BMC Cancer. 2016 Oct 21;16(1):816. doi: 10.1186/s12885-016-2856-2. PMID 27769214